CLINICAL TRIAL: NCT01586390
Title: Functional Treatment for Acute Ankle Sprains: Softcast Wrap Versus MOKcast. A Prospective Randomized Single-centre Trial
Brief Title: Functional Treatment for Acute Ankle Sprains: Softcast Wrap Versus MOKcast
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spaarne Gasthuis (Other)
Responsible Party: Principal Investigator, Daniel Mensch, MD, Spaarne Gasthuis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRAPvsMOK
Record Dates: First submitted 2012-04-23; First posted 2012-04-26 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Acute Ankle Sprain; Ankle Ligament Rupture; Ankle Injuries
Keywords: Ankle Sprain; Ankle Distortion; Functional treatment; Brace treatment
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MOK (Experimental): Adjustable and removable brace made out of Softcast material
  Interventions: Other: Ankle sprain treated with removable ankle support
- WRAP (Active Comparator): Softcast ankle cast
  Interventions: Other: Functional treatment for ankle sprain using ankle cast

INTERVENTIONS:
Other: Functional treatment for ankle sprain using ankle cast — Functional treatment for ankle sprain using ankle cast
  Arms: WRAP
Other: Ankle sprain treated with removable ankle support — Ankle sprain functionally treated with removable and adjustable ankle support
  Arms: MOK

SUMMARY:
In this study we compare two treatment options for ankle sprains. 100 patients were randomised between a flexible cast treatment and a removable and adjustable brace made out of the same materials.

Follow-up was 4 months. Primary outcome were functional scores. Secondary outcome measures were patient satisfaction scores with treatment as well as treatment result.

ELIGIBILITY:
Inclusion Criteria:

• Grade 2 and 3 acute ankle sprains

Exclusion Criteria:

* history of ankle sprains with persistent instability
* grade I lateral ankle sprains
* ankle fracture
* bilateral ankle sprains
* previous ankle ligament surgery
* neuromuscular disorders of the lower extremities
* rheumatoid arthritis,
* alcoholism,
* serious psychiatric or neurological illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Functional scores according to Karlsson score | Follow-up of 4 months
  The modified KSS gives a score from 0-90 on perceived function of the ankle and foot, divided over eight topics relevant to daily function. The modified KSS at 4 months was the primary endpoint.

SECONDARY OUTCOMES:
Pain | follow-up of 4 months
  Measured by Visual analogue scale (1-10)
Satisfaction score | follow-up of 4 months
  satisfaction scores with treatment as well as treatment result on scale 1-10

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Mensch, MD, Principal Investigator — Spaarne Gasthuis
Locations (1):
- Spaarneziekenhuis, Hoofddorp, Netherlands